CLINICAL TRIAL: NCT01217385
Title: Diffuse Optical Spectroscopy Imaging in Monitoring and Predicting Response in Patients With Locally Advanced Breast Cancer Undergoing Chemotherapy Before Surgery
Brief Title: Monitoring and Predicting Chemotherapy Response Using DOSI
Acronym: ACRIN6691
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000674337; ACRIN-6691 (Other: ACRIN Foundation); U01CA080098 (NIH); U01CA079778 (NIH)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Spectrometry, Mass, Matrix-Assisted Laser Desorption-Ionization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DOSI Pre-Surgery (Experimental): Participants undergo approximately four assessments of breast health using the DOSI technology during treatment and prior to surgery for breast cancer.
  Interventions: Procedure: DOSI

INTERVENTIONS:
Procedure: DOSI — Bedside DOSI images of the tissue concentrations of deoxy-hemoglobin (ctHHb), oxy-hemoglobin (ctHbO2), water (ctH2O), lipid, tissue oxygen saturation (StO2), and TOI (ctHHb x tH2O/lipid) were acquired on both breasts up to four times during neoadjuvant chemotherapy (NAC) treatment.
  Other Names: Diffuse Optical Spectroscopic Imaging; Laser spectroscopy; Optical Breast Imaging

SUMMARY:
RATIONALE: New imaging procedures, such as diffuse optical spectroscopy imaging, may help measure a patient's response and allow doctors to plan better treatment.

PURPOSE: This clinical trial studies diffuse optical spectroscopy imaging in monitoring and predicting response in patients with locally advanced breast cancer undergoing chemotherapy before surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether the percentage change in the diffuse optical spectroscopy imaging (DOSI) measurement of the tumor/normal (T/N) tissue optical index (TOI) from baseline to mid-therapy is predictive of the final pathologic response of the primary tumor in patients with locally advanced breast cancer treated with neoadjuvant chemotherapy.

Secondary

* To investigate whether change of TOI measurements from baseline to post-therapy are predictive of the final pathologic response in these patients treated with this regimen.
* To investigate whether baseline TOI measurements are associated with final pathologic response in patients treated with this regimen.
* To investigate whether TOI measurements at baseline, change from baseline to mid-therapy, and change from baseline to post-therapy correlate with available MRI volumetric imaging measurements.
* To investigate whether changes on TOI measurements from baseline to mid-therapy, and from baseline to post-therapy, correlate with other standard-of-care imaging and/or any MRI-imaging measurements.
* To explore whether additional optical endpoints and indices obtained during DOSI measurements can be used to predict final pathologic response in patients treated with this regimen.
* To determine a cutpoint for the percent change of TOI from baseline to mid-therapy that is predictive of pathological complete response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients undergo diffuse optical spectroscopy imaging (DOSI) at baseline, 5-10 days after initiation of neoadjuvant chemotherapy, during early- and mid-neoadjuvant therapy, and within 21 days after completion of neoadjuvant therapy. Results are compared to standard-of-care imaging (e.g., MRI, ultrasound, mammography). Patients then undergo surgery.

ELIGIBILITY:
Inclusion Criteria

1. Pathologically confirmed diagnosis of invasive breast cancer, determined to be a candidate for primary systemic (neoadjuvant) therapy and for surgical resection of residual primary tumor following completion of neoadjuvant therapy;
2. Tumor size >2cm, measured on imaging or estimated by physical exam;
3. No contraindications for primary chemotherapy;
4. Planned definitive breast surgery (mastectomy or lumpectomy/breast conservation) following completion of neoadjuvant therapy;
5. Age 18 years or older;
6. ECOG Performance Status ≤ 2 (Karnofsky ≥ 60%; see Appendix II);
7. Normal organ and marrow function as follows:

   * leukocytes ≥ 3,000/μl;
   * absolute neutrophil count ≥ 1,500/μl;
   * platelets ≥ 100,000/μl;
   * total bilirubin within normal institutional limits;
   * AST(SGOT)/ALT(SGPT) ≤ 2.5 times the institutional upper limit of normal;
   * creatinine within normal institutional limits; OR
   * creatinine clearance ≥ 30 mL/min/1.73 m2 for patients with creatinine levels above institutional normal;
8. If female, postmenopausal for a minimum of one year, OR surgically sterile, OR not pregnant, confirmed by a pregnancy test as per institutional Standard of Care (SOC), and willing to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation;
9. Able to understand and willing to sign a written informed consent document and a HIPAA authorization in accordance with institutional guidelines;

Exclusion Criteria

1. Previous treatment (chemotherapy, radiation, or surgery) to involved breast; including hormone therapy;
2. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements;
3. Medically unstable;
4. Under age 18;
5. Pregnant or nursing;
6. Previous malignancy, other than basal cell or squamous cell carcinoma of the skin or in situ carcinoma of the cervix, from which the patient has been disease free for less than 5 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2014-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J. Tromberg, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Irvine, California
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: Yes
See ACRIN data Sharing Policy:
  Monitoring and Predicting Breast Cancer Neoadjuvant Chemotherapy Response Using Diffuse Optical Spectroscopic Imaging (DOSI)
Time Frame: after publication of Primary manuscript
Access Criteria: See ACRIN data sharing policy
URL: https://www.acrin.org/RESEARCHERS/POLICIES/DATAANDIMAGESHARINGPOLICY.aspx

REFERENCES:
- [Result] Tromberg BJ, Butler JA, Mankoff DA, et al.: ACRIN 6691 monitoring and predicting breast cancer neoadjuvant chemotherapy response using diffuse optical spectroscopic imaging (DOSI). [Abstract] J Clin Oncol 29 (Suppl 15): A-TPS249, 2011.
- [Result] Tromberg BJ, Zhang Z, Leproux A, O'Sullivan TD, Cerussi AE, Carpenter PM, Mehta RS, Roblyer D, Yang W, Paulsen KD, Pogue BW, Jiang S, Kaufman PA, Yodh AG, Chung SH, Schnall M, Snyder BS, Hylton N, Boas DA, Carp SA, Isakoff SJ, Mankoff D; ACRIN 6691 investigators. Predicting Responses to Neoadjuvant Chemotherapy in Breast Cancer: ACRIN 6691 Trial of Diffuse Optical Spectroscopic Imaging. Cancer Res. 2016 Oct 15;76(20):5933-5944. doi: 10.1158/0008-5472.CAN-16-0346. Epub 2016 Aug 15. PMID 27527559
- See also: National Cancer Institute's clinical trials database — https://clinicaltrials.gov/ct2/show/NCT01217385

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven institutions were approved to enroll a total of 60 female breast cancer patients: Enrollment began in June 2011 and completed in June 2013. All institutions activated concurrently, except MD Anderson Cancer Center and Boston University, which joined the study in January and May 2013, respectively.
Groups:
- Diffuse Optical Spectroscopy Imaging (DOSI): Participants undergo approximately four assessments of breast health using the Diffuse optical spectroscopy imaging (DOSI)technology during treatment and prior to surgery for breast cancer.
  DOSI: Bedside DOSI images of the tissue concentrations of deoxy-hemoglobin (ctHHb), oxy-hemoglobin (ctHbO2), water (ctH2O), lipid, and TOI (ctHHb x tH2O/lipid) were acquired on both breasts up to four times during neoadjuvant chemotherapy (NAC) treatment.
Period: Overall Study
Arm/Group | Diffuse Optical Spectroscopy Imaging (DOSI)
Started | 60
Completed | 34
Not Completed | 26
Not completed — Withdrawal by Subject | 3
Not completed — DOSI not performed/not eval | 12
Not completed — Central Path not Available | 1
Not completed — Normal Breast TOI not available | 10

BASELINE CHARACTERISTICS:
Groups:
- Diffuse Optical Spectroscopy Imaging (DOSI): Participants undergo approximately four assessments of breast health using the DOSI technology during treatment and prior to surgery for breast cancer.
  DOSI: Bedside DOSI images of the tissue concentrations of deoxy-hemoglobin (ctHHb), oxy-hemoglobin (ctHbO2), water (ctH2O), lipid, and TOI (ctHHb x tH2O/lipid) were acquired on both breasts up to four times during neoadjuvant Chemotherapy (NAC) treatment.
Arm/Group | Diffuse Optical Spectroscopy Imaging (DOSI)
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 19
  More than one race | 0
  Unknown or Not Reported | 3
Histologic findings [Count of Participants; unit: Participants]
  Invasive (infiltrating) ductal carcinoma (IDC) | 16
  Invasive lobular carcinoma (ILC) | 3
  Ductal Carcinoma In Situ (DCIS)/ILC | 11
  IDC/ILC | 2
  Other/not available | 2
estrogen receptor (ER) status [Count of Participants; unit: Participants]
  Positive | 24
  Negative | 7
  Unknown | 3
progesterone receptor (PR) status [Count of Participants; unit: Participants]
  Positive | 19
  Negative | 12
  Unknown | 3
cell division marker (Ki67) status [Count of Participants; unit: Participants]
  Positive | 17
  Negative | 2
  Unknown | 15
hormone receptor 2 (Her2/neu) status from Immunohistochemistry (IHC): [Count of Participants; unit: Participants]
  0 - HER2-negative | 4
  1 - HER2-negative | 8
  2 - equivocal | 8
  3 - HER2-positive | 4
  unknown/not available | 10
fluorescence in situ hybridization (FISH) status [Count of Participants; unit: Participants]
  Amplified | 7
  Non amplified | 14
  Unknown/not available | 13
Areolar tumor [Count of Participants; unit: Participants]
  Areolar tumor | 17
  Nonareolar tumor | 17

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of %Change in TOI Between Baseline and Mid-therapy to Predict Pathologic Response (pCR +/-)
Description: This measure will look at the Accuracy of % change in DOSI measured Tumor Optical Index (TOI) from baseline to mid therapy to predict pathologic response (pCR+ v pCR-) Pathologic response (dichotomized into responders (pCR+) and non-responders (pCR-) based pathologic assessment) will be used as the reference standard and Accuracy will be determined using receiver operating characteristic (ROC) analysis to determine the ROC Area Under the Curve (AUC).
Time Frame: From baseline to mid-therapy
Population: Bedside DOSI images of the tissue concentrations of TOI (ctHHb x tH2O/lipid) acquired on both breasts at baseline and mid-therapy during neoadjuvant chemotherapy (NAC) treatment.
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- Diffuse Optical Spectroscopy Imaging (DOSI: Participants undergo approximately four assessments of breast health using the DOSI technology during treatment and prior to surgery for breast cancer.
  DOSI: Bedside DOSI images of the tissue concentrations of deoxy-hemoglobin (ctHHb), oxy-hemoglobin (ctHbO2), water (ctH2O), lipid, and TOI (ctHHb x tH2O/lipid) were acquired on both breasts up to four times during NAC treatment.
Arm/Group | Diffuse Optical Spectroscopy Imaging (DOSI
Number analyzed (Participants) | 34
probability | 0.60 [0.39 to 0.81]
Statistical Analysis 1: Comparison: Diffuse Optical Spectroscopy Imaging (DOSI; This analysis will look at the ability of the % change in DOSI measured tumor Optical Index (TOI) from baseline to mid-therapy to predict pathologic response using logistic regression. Pathologic response (dichotomized into responders and non-responders) will be used as the reference standard and %change in TOI ratio (dichotomized at -40%) will be used to estimate pCR (+/-)= alpha + beta1(%change TOI); Test type: Equivalence — under the NULL, it is assume that there is no difference between a 40% decrease in TOI, and a less than 40% decrease or an increase in TOI in their ability to predict pCR+; p = 0.059, Regression, Logistic — 5% alpha threshold for significance; Odds Ratio (OR) = 4.667, 95% CI 2-sided [0.95 to 23.04]

2. Secondary Outcome: %Change in TOI Between Baseline and Mid-therapy to Predict pCR+; Stratified by Progesterone Receptor (PR) Status (Positive, Negative, Unknown )
Description: Pathologic Complete response vs Non-Complete response, by PR status Progesterone Receptor Status (positive, negative, unknown ) is determined at pathological assessment of the tumor sample.
  %change in TOI is evaluated from baseline to mid-therapy.
Time Frame: baseline to mid-therapy
Population: Analysis population consists of the 34 participants with both baseline and mid-therapy TOI measurements.
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- PR+ Participants: Participants who are PR Positive (PR+)
- PR- Participants: Participants who are Progesterone Receptor Negative (PR-)
- PR? Participants: Participants whose PR status is unknown
Arm/Group | PR+ Participants | PR- Participants | PR? Participants
Number analyzed (Participants) | 19 | 12 | 3
percentage change | -29.874 (31.349) | -14.605 (107.425) | -45.701 (25.237)
Statistical Analysis 1: Comparison: PR+ Participants vs PR- Participants; The Null is that the odd ratio is the same in both the PR+ and PR- subjects fro the model including %change in TOI form baseline to mid-therapy (dichotomized at <=-40%), PR status (+/-) and the interaction between them; Test type: Equivalence — test for the equivalence of %change in TOI ratio (dichotomized at <=-40%), between PR+ and PR- groups, with interaction; p = 0.8193, Regression, Logistic — significance at alpha=0.05; p-value represents the interaction between %TOI (dichotomized at <=-40%), and PR status; Slope = 0.4463, Standard Error of Mean 1.953 — Multivariate logistic regression model using % change in TOI ratio (T/N) (baseline to mid-therapy) dichotomized at -40%, PR status, and the corresponding interaction

3. Secondary Outcome: Accuracy of %Change in TOI Between Baseline and Mid-therapy to Predict pCR+; Stratified by Oxygen Saturation (St02)
Description: subset analysis, subjects were stratified using the median tumor StO2
  %change TOI Between Baseline and Mid-therapy dichotomized at -40% stratified by the set evaluable subjects with baseline tumor StO2 dichotomized at 76.9%. (i.e. population median).
  Accuracy will be determined using ROC analysis to determine the ROC Area Under the Curve (AUC).
Time Frame: baseline to mid-therapy
Population: evaluable subjects with baseline tumor StO2 dichotomized at 76.9%. (i.e. population median) and %change TOI dichotomized at -40%
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- StO2 Negative: Evaluable subjects with measurable baseline tumor oxygen saturation StO2 <= 76.9%. (i.e. population median)
- StO2 Positive: Evaluable subjects with measurable baseline tumor oxygen saturation StO2 > 76.9%. (i.e. population median)
Arm/Group | StO2 Negative | StO2 Positive
Number analyzed (Participants) | 17 | 17
probability | 0.38 [0.08 to 0.68] | 0.83 [0.63 to 1]
Statistical Analysis 1: Comparison: StO2 Positive; Test type: Other; p = 0.043, Regression, Logistic; Odds Ratio (OR) = 16.5, 95% CI 2-sided [1.09 to 250.15]
Statistical Analysis 2: Comparison: StO2 Negative; Test type: Other; p = 0.406, Regression, Logistic; Odds Ratio (OR) = 2.86, 95% CI 2-sided [0.24 to 33.90]

4. Secondary Outcome: Estimate the Optimal Cutpoint for %Change in TOI From Baseline to Mid-therapy to Predict pCR
Description: Determine the optimal cutpoint (aka Youden-index) for %Change in TOI ratio (T/N) to maximize sensitivity and specificity in the predication of pCR
Time Frame: baseline to mid-therapy
Population: participants having TOI ratio (T/N) using tumor breast normal at baseline and mid-therapy and have pathologic response data.
Measure: Number; unit: percentage change in TOI
Arm/Group | Diffuse Optical Spectroscopy Imaging (DOSI)
Number analyzed (Participants) | 44
percentage change in TOI | -32.527

ADVERSE EVENTS:
Groups:
- DOSI: Participants undergo approximately four assessments of breast health using the DOSI technology during treatment and prior to surgery for breast cancer.
  DOSI: Bedside DOSI images of the tissue concentrations of deoxy-hemoglobin (ctHHb), oxy-hemoglobin (ctHbO2), water (ctH2O), lipid, and TOI (ctHHb x tH2O/lipid) were acquired on both breasts up to four times during NAC treatment.
Arm/Group | DOSI
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No